CLINICAL TRIAL: NCT06021366
Title: Treatment Patterns With Brolucizumab in Germany - a Retrospective Cohort Study Based on Longitudinal Prescription Data: REALIZE Study
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258A2015
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (8):
- 12-month follow-up cohort
- Treatment-naïve 12-month sub-cohort
- Treatment-experienced 12-month sub-cohort
- Treatment-experienced, persistent 12-month sub-cohort
- 18-month follow-up cohort
- Treatment-naïve 18-month sub-cohort
- Treatment-experienced 18-month sub-cohort
- Treatment-experienced, persistent 18-month sub-cohort

SUMMARY:
REALIZE was a single-arm retrospective cohort study which described treatment patterns with brolucizumab, including treatment intervals between anti-vascular endothelial growth factor (VEGF) injections before and after a switch to brolucizumab.

This study was conducted using German patient-level prescription data and the prescription date was used as a proxy for anti-VEGF injection date.

The study period was defined from the date of the first available anti-VEGF injection in the dataset to 30 November 2021. The index date for each patient was the date of the first brolucizumab injection, which could be anytime between 01 March 2020 (since brolucizumab became available in Germany for use outside of clinical trials in March 2020) and 30 November 2021. The date of the patient's first neovascular age-related macular degeneration (nAMD) diagnosis was assumed to be the date of the first anti-VEGF prescription in the database for that patient, from January 2015 onwards.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged ≥50 years with a nAMD diagnosis, who received ≥1 brolucizumab prescription regardless of prior anti-VEGF treatment, and had a minimum of 12-month follow-up from index date.

Exclusion Criteria:

* Patients without a record of prescription of any drug in the six months before the index date (pre-index period).
* Patients with evidence of bilateral treatment with brolucizumab.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 2089 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Number of brolucizumab injections | Up to 12 months

SECONDARY OUTCOMES:
Time difference between the last anti-VEGF treatment interval before switch to brolucizumab and the last brolucizumab treatment interval at 12 months | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Porto Salvo, Portugal